CLINICAL TRIAL: NCT00004347
Title: The Effects of Dietary Cholesterol in the Smith-Lemli-Opitz Syndrome
Brief Title: Phase II Study of Dietary Cholesterol for Smith-Lemli-Opitz Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00334-0068; OHSU-4019
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: Smith-Lemli-Opitz syndrome; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Genetic Diseases, Inborn; Rare Diseases | interventions — Diet

INTERVENTIONS:
Behavioral: diet

SUMMARY:
OBJECTIVES: I. Examine the intestinal absorption of dietary cholesterol in patients with Smith-Lemli-Opitz syndrome.

II. Measure the effect of dietary cholesterol on plasma sterol composition. III. Quantify basal cholesterol synthesis, turnover of cholesterol and 7-dehydrocholesterol, and the effects of dietary cholesterol on these parameters.

IV. Identify fecal bile acid excretion quantitatively and qualitatively in these patients.

V. Compare the incorporation of deuterated water into plasma cholesterol, 7-dehydrocholesterol, and other intermediates, and assess the effect of dietary cholesterol on this incorporation.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are treated with 2 dietary regimens for 1 to 3 weeks: high cholesterol and cholesterol-free. Cholesterol is provided in the form of egg yolk. The absorption and metabolism of cholesterol are evaluated with plasma and fecal studies. Deuterated water is given to patients followed by analysis of deuterium in plasma cholesterol and other intermediates, including 7-dehydrocholesterol.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Smith-Lemli-Opitz syndrome

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1995-11

CONTACTS AND LOCATIONS:
Overall Officials: William Connor, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States